CLINICAL TRIAL: NCT02510846
Title: Impact of an Intensive Multimodal Educative Program on Behavioral Disorders of Patients With Profound Multiple Disabilities and on the Quality of Life and Feelings of Caregivers
Acronym: TDCHandi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: K140701; PHRIP140325 (Other: Assistance publique)
Record Dates: First submitted 2015-07-13; First posted 2015-07-29 (Estimated); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Polyhandicap; Behavior Disorders
Keywords: Polyhandicap; Behavior disorders; Educative program; Caregivers; Quality of life.
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intensive educative program (Experimental): 5 hours a week
  Interventions: Behavioral: Intensive educative management
- Usual practice of educative program (Active Comparator): 1 hour a week
  Interventions: Behavioral: Intensive educative management

INTERVENTIONS:
Behavioral: Intensive educative management — 5 hours a week

SUMMARY:
Profound multiple disabilities also called in French polyhandicap are defined by the combination of a deep mental disability and severe motor deficit with extreme restriction of autonomy. Life in institution for people with profound multiple disabilities induces emotional and educative deficiency and often conducts to behavioral disorders. These behavioral disorders also impact on quality of life and feelings of caregivers. An intensive multimodal educative program proposed to patients with profound multiple disabilities can improve their psychic well-being, reduce chronic pain and improve also quality of life and feelings of caregivers. The intensive multimodal educative program will be compared to the usual practice of educative program.

DETAILED DESCRIPTION:
People with profound multiples disabilities needs particular follow-up with education, care, communication and socialization.

Our hypothesis is that an intensive multimodal educative program of 5 hours a week during 12 months compared to the usual practice of 1 hour a week conducts to the reduction of behavioral disorders and improves the quality of life and feelings of caregivers.

This study is multicenter, controlled, randomized in two parallel groups and open-labelled comparing usual practice of educative program and intensive educative program during 12 months.

The evolution of predominant behavioral disorder and quality of life and feelings of caregivers is evaluated at inclusion (M0), six months after (M6) and twelve months after (M12).

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patient
* Age between 3 and 35 years old
* Patient with multiple disabilities defined by the following 5 criteria:

  1. reached or causal brain injury occurred before 3 years and
  2. profound mental disability (IQ lower than 35 or not assessable by psychometric tests when patients are too deficient) and
  3. motor disability (para-quadraparesis, hemiparesis, diplegia, ataxia, extrapyramidal motor disorders, neuromuscular disorders) and
  4. reduced mobility ( Gross Motor Function Classification System score: GMFCS III à V) and
  5. extreme autonomy restriction (FMI Functional Independency lower than 50)
* Patient with at least once per week of the following behavioral disorders:

  * Restlessness episodes (refusal of physical or verbal contact expressed by gestures aiming to push off other patients or caregivers and/or shouts when caregivers try to approach).

or

• Unexplained crying: according to the Riccilo S.C, Watterson T [Riccilo 1984] definition: fully or partially closed eyes, facial grim/wince and vocalization with or without tears.

or

* Rumination or
* Bruxism or
* Self-mutilations or
* Heteroagressif behavior (bite, pinch, hit) or
* Gestural stereotypies or
* Rythmic movements or
* Iterative frictions

Exclusion Criteria:

* No agreement of participation to the study by the holders of parental authority / legal guardian.

Ages: 3 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 63 (Actual)
Dates: Start 2016-01-15 (Actual); Primary Completion 2017-07-27 (Actual); Study Completion 2017-07-27 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy at 12 months of intensive multimodalitaire educational care compared to usual educational care of patients with multiple disabilities on behavioral disorders. | At the inclusion and 12 months
  The average number of predominant behavioral disorder will be evaluated by caregivers filling a form twice a day during 7 days.
  The predominant behavioral disorder will be identified by the caregivers after 15 days of observation among the following disorders:
  * Restlessness episodes
  * Unexplained crying
  * Rumination
  * Bruxism
  * Self-mutilations
  * Heteroagressif behavior
  * Gestural Stereotypies
  * Rythmic movements (swings)
  * Iterative friction

SECONDARY OUTCOMES:
Chronic pain. (EDSS scale) | At the inclusion, 6 months and 12 months.
  Pain evaluation with the validated EDSS scale
Evolution of frequency of behavior disorders. | At the inclusion, 6 months and 12 months.
  The behavioral disorders will be evaluated during 7 days with a form filled out twice a day by caregivers.
Consumption of psychotropic treatments. | At the inclusion and 12 months.
  Reduction of the number and/or dose of psychotropic treatments.
Evaluation of the impact of an intensive educative program for patients on chronic stress consequences on referent caregivers at the inclusion, 6 months and 12 months evaluated by the Maslach Burnout Inventory (MBI). | At the inclusion, 6 months and 12 months
Evaluation of the impact of an intensive educative program for patients on implemented strategy to deal with stress among referent caregivers at the inclusion and 12 months. with the Brief-COPE questionnaire. | At the inclusion and 12 months.
Evaluation of the impact of an intensive educative program for patients on emotional distress of referent caregivers evaluated at the inclusion and 12 months with the Hospital Anxiety and Depression Scale (HADS). | At the inclusion and 12 months
Evaluation of the impact of an intensive educative program for patients on quality of life of referent caregivers evaluated at the inclusion and 12 months with the WOQOL-Bref scale. | At the inclusion and 12 months
Evaluation of the impact an intensive educative program on the duration of behavioural problems by the average difference between the inclusion and at 12 months | At the inclusion and 12 months
Evaluation of the impact an intensive educative program on the disorder most invasive behaviour for the patient by the frequency of disappearance between the inclusion and at 12 months and the most pervasive disorder | At the inclusion and 12 months
  The most pervasive disorder is defined as the most harmful disorder for the patient and/or its management, according to the care teams responsible for each patient

CONTACTS AND LOCATIONS:
Overall Officials: Etienne GUILLUY, GUILLUY, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital La Roche Guyon, La Roche-Guyon, France